CLINICAL TRIAL: NCT00141895
Title: A Randomized Trial of Two Regimens of Misoprostol for Second Trimester Intrauterine Fetal Death
Brief Title: A Randomized Trial of Two Regimens of Misoprostol for Second Trimester Termination for Intrauterine Fetal Death
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Anwar Nassar, professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OGY.AN.03
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Labor Induction
Keywords: Intrauterine fetal death, 2nd trimester, induction
MeSH Terms: conditions — Stillbirth | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Vaginal Cytotec at doses of 400 microgram every 4 hours until delivery
  Interventions: Drug: Misoprostol
- B (Active Comparator): Sublingual Cytotec at doses of 400 microgram every 4 hours until delivery
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 2 tablets 200 micrograms Vaginal route
  Other Names: Cytotec
  Arms: A
Drug: Misoprostol — 2 tablets of 200 micrograms Sublingual route
  Other Names: Cytotec
  Arms: B

SUMMARY:
Misoprostol (Cytotec®) is a synthetic prostaglandin E1 analog that has been marketed in the United States since 1988 as a gastric cytoprotective agent. Despite a focused campaign by the manufacturer to curtail its use in obstetric practice, misoprostol has, over the past several years, gained widespread acceptance to effect the medical termination of pregnancy in the second trimester, either alone or after pretreatment with mifepristone. The primary reasons for this prompt incorporation into standard practice include its low cost and the lack of stringent storage requirements.

Vaginal administration seems to be more efficacious than when given orally. The use of sublingual misoprostol for first trimester abortions has been extensively investigated as evidenced by the large number of publications comparing sublingual to other routes of misoprostol for first trimester pregnancy termination, on the assumption that the sublingual route would have a similar efficacy of the vaginal route. In addition, the sublingual route would combine an easier administration with the added advantage of no restriction of mobility after administration. There has been no previous report in the literature comparing the use of misoprostol given sublingually to that given vaginally for the second trimester termination following intrauterine fetal death. Our aim is to compare efficacy, safety and patient satisfaction with misoprostol given vaginally (the current standard) to that given sublingually.

DETAILED DESCRIPTION:
Prostaglandins have been recognized as effective abortifacients for several decades. Misoprostol, a synthetic analogue of prostaglandin E1, has several advantages over other prostaglandins that include low cost, easy storage at room temperature, and favorable side effect profile. In recent years, misoprostol has attracted attention as an effective and cost-efficient agent for the medical interruption of the second-trimester pregnancy. Nowadays, misoprostol has been accepted widely as a safe and effective agent for labor induction during the second trimester. Various doses, routes, and protocols for medical termination of pregnancy during the second trimester have been investigated. The optimal dosage and route of administration, however, have yet to be defined. Previous studies have demonstrated greater efficacy with vaginal misoprostol versus oral administration in effecting mid-trimester termination. However, oral administration of any medication is preferred by patients and health care providers alike. The higher efficacy after vaginal administration may be explained by the pharmacokinetics of the drug. Zeiman et al showed that the systemic bioavailability of vaginally administered misoprostol is 3 times higher than that after oral administration. Plasma concentrations of its metabolite, misoprostol acid, peak one to two hours after vaginal application as compared with the peak seen 30 minutes following oral administration, and although peak levels are lower with the vaginal route, they are sustained longer and overall exposure to the drug is increased, perhaps because of the presystemic gastrointestinal or hepatic metabolism that occurs with the oral route. An additional explanation for the higher efficacy could be that there is a direct effect on the cervix that initiates the physiologic events that lead to increased uterine contractility. The sublingual route of administration has not been reported in the literature prior to 2001. Since then and partly because of issues relating to patient preference, investigators started studying the sublingual route of administration of misoprostol. In theory, the sublingual route could mimic vaginal administration pharmacokinetically, although there have been no such reported studies on this route of administration.

Although many studies have been published on the use of sublingual misoprostol for medical abortion in the first trimester, none were done to compare sublingual and vaginal routes in the case of second trimester termination for intrauterine fetal death. The 400-µg dose was chosen because it is the dose most commonly used orally and vaginally in various studies reported in the literature.

To the best of our knowledge, no study comparing sublingual to vaginal misoprostol for termination of pregnancy for intrauterine fetal death in the second trimester has been previously published in the literature. Therefore, this study, when completed will provide evidence on the relative effect and safety profile of different routes of administration of misoprostol for indicated second trimester termination.

The aim of our study is to compare the efficacy of a 400-µg sublingual dose of misoprostol Cytotec® (Searle Pharmaceuticals, Bucks, United Kingdom) administered at 4-hour intervals with an equivalent dose regimen administered vaginally in women admitted for second trimester termination for intrauterine fetal death. In addition, we want to assess patient acceptability of the 2 modes of administration.

The study hypothesis is that the sublingual route of administration of misoprostol is as effective as the vaginal route for induction of labor for mid trimester termination and is more acceptable to patients as compared to vaginal misoprostol.

Randomization procedure:

The randomization to vaginal or sublingual misoprostol will be based on a computer-generated table with the allocation concealed in sealed, sequentially numbered, brown envelopes, which had been prepared by the principal investigator that will not be involved in the clinical care of the patients. Because of the nature of the misoprostol administration, the patients and staff will not blinded to the randomization allocation.

Routine studies and procedures:

* A pelvic exam will be done to make sure that the patient is eligible for inclusion in the study (Bishop's score <8).
* Maternal pulse, blood pressure, and temperature will be recorded every 4 hours ( at the time of the insertion of the Misoprostol).
* After delivery of the fetus, all patients will receive 20 units of oxytocin in 1000 mL of intravenous crystalloid at an infusion rate of 125 mL per hour.
* Postpartum curettage will be performed at the discretion of the physician if the placenta had not delivered spontaneously 2 hours after the delivery of the fetus.
* Patients will receive intravenous narcotics or epidural anesthesia as needed for pain control.
* Antiemetics, antipyretics, and anxiolytics will be administered as indicated. Interventions: The women will give a full informed consent, after which they will be randomized to receive 400 µg of vaginal or sublingual misoprostol Cytotec® (Searle Pharmaceuticals, Bucks, United Kingdom) after admission to the induction ward. This dose and route of administration will be repeated every 4 hours, if required as long as the patient is undelivered up to 48 hours following initiation of induction.

The induction will be categorized as having failed if the woman was undelivered after 48 hours and then she would receive extraamniotic PGF2 instillation or high-concentration intravenous oxytocin, depending on their cervical status and amniotic membrane integrity. Another option would be a further attempt at cervical ripening with vaginal Prostin tablets (Upjohn Pharmaceuticals) after an interval of at least four hours following the last dose of misoprostol.

- The women will complete a brief questionnaire using a visual analogue scale to ascertain their perceptions of the process in terms of pain, control, and overall opinion of the procedure every 12 hours. The women will perform the pain scale assessments with a visual analogue ruler scaled from 0 to 10, with 0 representing no perception of pain and 10 representing the most intense pain ever experienced.

Statistical analysis Statistical analysis will be performed using the SPSS statistical package. Categoric data like maternal characteristics will be compared using Chi square when sample sizes support the approximation. Otherwise, categorical data will be analyzed with two-tailed Fisher exact test if the expected cell frequencies were small. Continuous variables will be compared by Student t test if assumptions of normality and homogeneity of variances appeared to be reasonable. Unpaired variables and differences in distributions will be compared using the Mann-Whitney test. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 14 and 24 weeks of gestation
* Both nulliparous and multiparous women
* An unfavorable cervix (Bishop's score less than 8)

Exclusion Criteria:

* Known contraindications to the use of prostaglandins (e.g. asthma)
* Previous uterine scar (previous cesarean or myomectomy where the endometrial cavity was entered)

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2004-09; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
-The main outcome measures will be the induction time, defined as the time from placement of the first dose of misoprostol until the time of delivery of the fetus. | 48 hours

SECONDARY OUTCOMES:
The entry characteristics of the patients, including age, height, weight, parity, gestational age at induction, indication for the induction, and cervical score before the start of the induction | 48 hours
The delivery rate within 24 hours of prostaglandin commencement | 48 hours
Number of doses of misoprostol given | 48 hours
Number of unsuccessful inductions | 48 hours
Length of hospital stay | 48 hours
Need for surgical intervention to remove the placenta | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anwar H Nassar, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352